CLINICAL TRIAL: NCT06225089
Title: Effect of Pericapsular Nerve Block on the Quality of Recovery After Shoulder Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Muhammed Halit Satici, Specialist, the member of department of Anesthesiology, Konya City Hospital, M.D, Konya City Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: pericapsüler nerve block
Record Dates: First submitted 2023-12-09; First posted 2024-01-25 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): All patients will receive routine monitoring ( ECG monitoring, SpO2, noninvasive blood pressure, and EtCO2) and routine anesthesia management. 20 gauge to patients IV Cannulation will be provided and isotonic fluid will be started according to the fluid calculation. General anesthesia induction 1mg midazolam IV, 2 mg/kg propofol IV, 1.5 mcg /kg fentanyl IV, 0.6 mg/kg rocuronium It will be done by giving IV. Patients will be intubated and the minimum amount of anesthesia required for maintenance alveolar Sevoflurane + 50% oxygen + 50% air will be given so that the concentration (MAC) value is 1 and 0.05 mcg/kg/min. remifentanil infusion will begin. The patients will then be released to the surgical team. After the surgical procedure is completed, all patients are given IV paracetamol 1 g 3x1, IV tenoxicam 20 mg 2x1, and IV dexamethasone 8mg will be administered 1x1. All patients will be administered IV 1mg/kg tramadol as rescue analgesic when NRS is 3 or above
- pericapsuler nerve block group (Active Comparator): all patients are given IV paracetamol 1 g 3x1, iv tenoxicam 20 mg 2x1, and IV dexmethasone 8mg will be administered 1x1. Patients in Group P will also receive a pericapsuler nerve block. All patients will be administered IV 1mg/kg tramadol as rescue analgesic when NRS is 3 or above. 4mg IV to all patients with nausea and vomiting Ondansetron will be administered. Once patients are extubated, they will be transferred to the postanesthetic care unit (PACU) for observation.
  Interventions: Drug: pericapsuler nerve block

INTERVENTIONS:
Drug: pericapsuler nerve block — -Ultrasound Guided pericapsuler nerve block: will be externally rotated and abducted to 45 degrees. The shoulder area will be sterilized with povidone-iodine. High-frequency linear ultrasound perpendicularly between the coracoid and the humeral head probe. The deltoid muscle, subscapular muscle and tendon, and humeral head will be identified on the ultrasound screen. With the in-plane technique, a 22 gauge, 50 millimeter (mm) simplex A peripheral nerve block needle will be used. After passing the deltoid muscle, the needle will contact the tendon of the subscapularis muscle. The needle will be slightly withdrawn and directed between the deltoid muscle and the tendon of the subscapularis muscle and a local injection consisting of will be applied.
  Arms: pericapsuler nerve block group

SUMMARY:
Shoulder arthroscopy surgery is one of the most common orthopedic surgical procedures. Participants experience severe pain after shoulder arthroscopy surgery. This causes the use of high amounts of opioids, delays healing, causes bleeding in the surgical area, and can cause physiological disorders by increasing the stress response. Multiple studies have been conducted for analgesic purposes in shoulder surgery. Tran et al., posterior to the glenohumeral joint of the superior part of the suprascapular nerve, posterior inferior part of the posterior branch of the axillary nerve, anterior superior part of subscapularis superior branch, anterior claimed that the axillary nerve innervates the inferior part. In their case report, reported that the pericapsular nerve block (PENG) applied to participants undergoing shoulder surgery provided postoperative analgesia for 16-24 hours pericapsuler nerve block, which is generally applied in hip surgeries, can be applied in shoulder surgery, but there is no large-scale study on pericapsuler nerve block in shoulder surgery, and there is still unknown whether there is a relationship between the pericapsuler nerve block to be applied and the quality of postoperative recovery. Recovery after surgery and anesthesia is complex.

DETAILED DESCRIPTION:
Shoulder arthroscopy surgery is one of the most common orthopedic surgical procedures. Participants experience severe pain after shoulder arthroscopy surgery. This causes the use of high amounts of opioids, delays healing, causes bleeding in the surgical area, and can cause physiological disorders by increasing the stress response. Multiple studies have been conducted for analgesic purposes in shoulder surgery. The axillary nerve is said to supply nerves to the inferior part of the suprascapular nerve, the posterior inferior part of the posterior branch of the axillary nerve, and the anterior superior part of the subscapularis superior branch. The study was done posterior to the glenohumeral joint. In their case report reported that the pericapsular nerve block (PENG) applied to participants undergoing shoulder surgery provided postoperative analgesia for 16-24 hours. The block, which is generally applied in hip surgeries, can be applied in shoulder surgery, but there is no large-scale study on the pericapsuler nerve block in shoulder surgery, and still unknown whether there is a relationship between the pericapsuler nerve block applied and the quality of postoperative recovery. Recovery after surgery and anesthesia is complex.

Application of the pericapsuler nerve block will provide better postoperative recovery and recovery scores in participants who will undergo shoulder arthroscopy surgery. The primary aim of this study is to evaluate the effectiveness of pericapsuler nerve block on postoperative recovery and recovery quality after shoulder arthroscopy surgery using the quality of recovery-15 questionnaire.

The secondery aim this study is to postoperatively immobilize and move numeric rating scale in participants undergoing shoulder arthroscopy surgery in which pericapsuler nerve block will be applied, the number of participants needing first-rescue analgesia, the time to first-rescue analgesia, and postoperative To evaluate complications, the number of patients in need of antiemetics, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will have unilateral shoulder arthroscopy
* Patients who will receive general anesthesia
* Patients aged 18-65
* Patients with ASAI-III
* in the hospital for at least 24 hours postoperatively

Exclusion Criteria:

* Patients who do not want to give consent
* Patients for whom regional anesthesia is contraindicated
* Patients with ASA IV and above
* Patients with confusion
* Patients with a bad bleeding profile using anticoagulants
* Patients with infection in the area to be treated
* Emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
quality of recovery-15T | One day
  The primary evaluation criteria will be the recording of Quality of recovery-15 scores, which indicate the quality of recovery of patients before and 24 hours after surgery. QoR = -15 (0-150; 0 = lowest degree of satisfaction, 150 = highest degree of satisfaction).

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No